CLINICAL TRIAL: NCT00777166
Title: Phase 4 Study of Oxytocin Used During Cesarean Section
Brief Title: Cardiac Effects of Oxytocin Administrated During Cesarean Section, Signs of Myocardial Ischemia
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Uppsala University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Single Group | Masking: Triple | Purpose: Treatment
Other Study IDs: 2004-004929-99
Record Dates: First submitted 2008-10-21; First posted 2008-10-22 (Estimated); Last update posted 2014-03-14 (Estimated); Status verified 2014-03

CONDITIONS: Myocardial Ischemia; Hypotension; Bloodloss
Keywords: oxytocin; ST depression; cesarean section; blood loss
MeSH Terms: conditions — Myocardial Ischemia; Hypotension; Hemorrhage | interventions — Oxytocin

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator
Oversight: Data Monitoring Committee: No

ARMS (2):
- 1 (Active Comparator): oxytocin 5 units
  Interventions: Drug: oxytocin
- 2 (Active Comparator): oxytocin, 10 units
  Interventions: Drug: oxytocin

INTERVENTIONS:
Drug: oxytocin — oxytocin 5 units diluted with normal saline to a total volume of 10 mL
  Other Names: syntocinon; Pitcotin
  Arms: 1
Drug: oxytocin — oxytocin 10 units diluted with normal saline to at total volume of 10 mL.
  Other Names: Syntocinon; Pitcotin
  Arms: 2

SUMMARY:
Oxytocin has cardio vascular effects as hypotension, tachycardia and possibly coronary spasm. The uterotonic effect of the drug is used during cesarean section, to minimize blood loss.ECG changes suggestive of cardiac ischemia (ST depression) has been showed in previous studies of patients undergoing cesarean section i regional anaesthesia. The effect of oxytocin on this outcome has not been investigated to any extent.

In the current study, we tested the hypothesis that there was no difference in occurrence of ECG changes (ST segment depression) between two doses of oxytocin. Participants were randomized to receive either 5 or 10 units of oxytocin in a double blinded fashion.

Main outcome measure is occurrence of significant ST depression on ECG. Secondary outcome measures are mean arterial pressure, heart rate, blood loss, symptoms as chest pain, shortness of breath and feeling of heaviness on the chest.

DETAILED DESCRIPTION:
All healthy term participants scheduled to undergo elective caesarean section under spinal anaesthesia at the Department of Obstetrics and Gynecology, University Hospital, Uppsala Sweden and who were > 18 years old, were candidates for inclusion in the study. .

The study was approved by the regional ethics committee and informed written consent was obtained from each participant.

ECGs were recorded by continuous ambulatory ECG (Holter) monitoring (GE Medical systems SEER/MARS, UK) during the peroperative period utilizing leads V3, V5 and avF. As secondary outcomes, symptoms as chest pain, shortness of breath and feeling of heaviness on the chest and, Troponin I levels 12 hours postoperatively, were recorded. Also, as secondary outcomes, differences in blood pressure, heart rate, and blood loss were measured.

Before induction of anaesthesia, patients received 1000 mL of lactated Ringer's solution intravenously. Thereafter an additional 500-1000 mL of lactated Ringer's solution or 500 mL Hydroxyethyl starch was infused if considered needed by the anaesthesiologist.

Spinal anaesthesia was established in the sitting position at lumbal interspace L2/L3 or L3/L4. Non invasive blood pressure (systolic, diastolic and mean arterial pressure, MAP) and heart rate was monitored every 2 minutes, throughout surgery. Oxytocin was given as an intravenous bolus dose immediately after clamping of the umbilical cord. Blood loss during the operation was estimated and recorded. During surgery, any spontaneous complaints by the patients of symptoms as chest pain, shortness of breath and feeling of heaviness on the chest, was recorded as well as duration of symptoms. Episodes of chest pain were assessed with the visual analogue scale (VAS).

Troponin I, as a marker of ischemic myocardial damage, was sampled 12 hours postoperatively.

The incidence of ECG changes related to different doses of intravenous bolus doses of oxytocin (5 and 10 units) during caesarean section is unknown. In a pilot study preceding the present study, 5 units oxytocin were administrated and the incidence of ECG changes was 15%. With the assumption that ECG changes could occur in 50% of subjects receiving 10 units oxytocin and based on 0.8 power to detect a significant difference (P = 0.05, two-sided), 25 patients were required for each study group. An interim analysis performed after inclusion of 50 patients revealed that ECG-changes occured in 8 and 24 % respectively in the two groups of 5 and 10 units of oxytocin. An additional 50 patients were allocated and a second interim analysis planned.

A computer-generated randomisation list with block of four was drawn up by a statistician and given to the pharmacy department who performed the randomisation. The procedure ensured allocation concealment.

All participants, health care providers, investigators and other persons (cardiologist) were blinded to treatment assignment for the duration of the study.

The Statistical Package for Social Sciences (SPSS) for Windows, version 15.0, was used (SPSS, Inc., Chicago, IL, USA). To compare group distributions the chi-squared test or Fisher's exact test was applied and the Mann-Whitney U-test or t-test for continuous variables. A p-value < 0.05 was considered to indicate a significant difference

ELIGIBILITY:
Inclusion Criteria:

* Healthy women >/= 18 years scheduled to planned cesarean section

Exclusion Criteria:

* BMI > 35
* Multiple birth
* Complications to pregnancy
* Non proficiency in the Swedish language

Ages: 18 Years to 45 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 103 (Actual)
Dates: Start 2005-12; Primary Completion 2008-07 (Actual); Study Completion 2008-07 (Actual)

PRIMARY OUTCOMES:
ST segment depression on ECG | 30 minutes

SECONDARY OUTCOMES:
mean arterial blood pressure, heart rate, blood loss and symptoms as chest pain | 60 minutes

CONTACTS AND LOCATIONS:
Overall Officials: Ove Axelsson, Professor, Principal Investigator — Uppsala University, Sweden
Locations (1):
- University hospital Uppsala, Uppsala, Sweden